CLINICAL TRIAL: NCT04203966
Title: Mental Health and Well-being of People Who Seek Help From Their Member of Parliament
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: HR-16/17-3220
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2019-12

CONDITIONS: Common Mental Disorders; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Common mental disorders/ versus no common mental disorders: No intervention This is a prevalence study- presence of common mental disorders (CMDs) will be assessed using the 12-item general Health Questionnaire, with responses above validated cut-points taken to indicate presence of CMDs
  Interventions: Diagnostic Test: 12-item General Health Questionnaire (GHQ-12)
- Alcohol use disorders/ versus no alcohol use disorders: No intervention This is a prevalence study- presence of alcohol use disorders will be assessed using the World Health Organization (WHO) AUDIT, with responses above validated cutpoints taken to indicate presence of alcohol use disorders
  Interventions: Diagnostic Test: WHO AUDIT (World Health Organization- Alcohol Use Disorders Inventory Tool)

INTERVENTIONS:
Diagnostic Test: 12-item General Health Questionnaire (GHQ-12) — Structured validated screening tools to assess for the presence of CMDs, administered to participants who have consented to take part in the study by completing responses either via survey monkey, or if they prefer through paper questionnaires posted to them
  Groups: Common mental disorders/ versus no common mental disorders
Diagnostic Test: WHO AUDIT (World Health Organization- Alcohol Use Disorders Inventory Tool) — Structured validated screening tools to assess for the presence of alcohol use disorders, administered to participants who have consented to take part in the study by completing responses either via survey monkey, or if they prefer through paper questionnaires posted to them
  Groups: Alcohol use disorders/ versus no alcohol use disorders

SUMMARY:
This is an observational study to assess the prevalence of common mental disorders and alcohol use disorders in a population of individuals seeking help from their Member of Parliament (MP) in the UK.

DETAILED DESCRIPTION:
Members of Parliament (MP) in the United Kingdom (UK) represent the interests of their constituents. Constituents may contact their MP for assistance if they feel that they have been treated unfairly by a government department or agency, have concerns relating to their local area, or are wanting support from their MP for a campaign they are involved in. In order to fulfil their duty to constituents, MPs hold regular surgeries which allow anyone with a concern to meet with them to discuss the issue in question further. Given the role of the MP in representing people who may be in the midst of stressful events, such as a dispute, it is possible that mental health problems may be more prevalent in this population. However, at present MPs are not given any additional training in recognising mental distress, and may not know how to appropriately sign-post people to appropriate supportive services, nor do MPs receive advice in supporting such individuals. To the best of the investigator's knowledge, there have been no prior studies in this area. The findings of this study will inform initiatives to improve MP working practices, to and raise awareness of the mental health challenges faced by their constituents, with the aim of better meeting the mental health needs of constituents who attend MP surgeries in the future.

ELIGIBILITY:
Inclusion Criteria:

* Attending selected MP surgeries (e.g. in Central Suffolk & North Ipswich)
* Over the age of 18
* Must be able to complete paper or online questionnaires.
* Have consented to take part in the study

Exclusion Criteria:

- Unable to complete questionnaires on their own/ unaided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People seeking help from their MP over study collection period
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Presence of common mental disorders indicated by scores above validated cutpoints on the GHQ-12 | Cross-sectional analysis, data was collected from September 2018, with exposures and outcomes collected at the same time points (ie. when people fill out the questionnaire). Time frame for analysis will be through to study completion.
  The 12-item General Health Questionnaire (GHQ-12) is a structured validated screening tool to assess for the presence of CMDs, administered to participants who have consented to take part in the study by completing responses either via survey monkey, or if they prefer through paper questionnaires posted to them. We will use validated cut points, individuals scoring above these (for example 4 or more on the GHQ-12) will be determined as having a common mental disorder

SECONDARY OUTCOMES:
Presence of alcohol use disorders, indicated by scores above validated cutpoints on the WHO AUDIT tool | Cross-sectional analysis, data was collected from September 2018, with exposures and outcomes collected at the same time points (ie. when people fill out the questionnaire). Time frame for analysis will be through to study completion.
  The World Health Organization (WHO) AUDIT is a structured validated screening tool to assess for the presence of alcohol use disorders, administered to participants who have consented to take part in the study by completing responses either via survey monkey, or if they prefer through paper questionnaires posted to them. We will use validated cutpoints to assess for the presence of harmful and hazardous alcohol use disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- IoPPN, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No